CLINICAL TRIAL: NCT05298579
Title: Comparison of the Efficiency of Yoga Exercises Applied With Two Different Technological Access in White Collar Employees
Brief Title: Yoga Exercises Applied With Two Different Technological Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc.Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BiruniA
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Work Related Stress; Pain; Fatigue
Keywords: white collar workers; yoga; remote exercise
MeSH Terms: conditions — Occupational Stress; Pain; Fatigue

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessors will be blind to the group allocation. The investigators will be blind to the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Yoga exercises applied by video-conference method accompanied by a physiotherapist.
  Evaluations and yoga exercises will be applied to the participants in this group through the "Zoom program". Yoga exercises were created with reference to studies in the literature. It will be applied for 8 weeks, 3 days a week and 40-45 minutes, at a time determined jointly by the physiotherapist and the participant (Table 1). Before starting the program, an informative broadcast will be made to the participants and groups of 6-8 people will be formed.
  Interventions: Other: Yoga exercises
- Group B (Active Comparator): Yoga exercises performed asynchronously accompanied by videos. Exercise videos will be broadcast to the participants in this group through the "YouTube program". The shooting of the exercise videos will be completed in advance and uploaded to a channel opened on YouTube. All posts made in this channel will only be open to individuals participating in the research during the duration of the study. Yoga exercises were created with reference to studies in the literature. It will be applied for 8 weeks, 3 days a week and 40-45 minutes. Participants will be able to access the exercise videos at a time they want (Table 2). Participants will be encouraged to achieve weekly targeted training sessions and to keep an exercise diary.
  Interventions: Other: Yoga exercises

INTERVENTIONS:
Other: Yoga exercises — Yoga-based exercise training includes a warm-up and cool-down period for beginners

SUMMARY:
Yoga, a form of exercise designed to bring balance and health to the physical, mental, emotional and spiritual dimensions of the individual, will benefit many white-collar workers by using popular technological environments to increase overall physical activity and well-being. The aim of this study is to examine the effects of yoga exercises applied with two different technological access in white-collar employees on musculoskeletal pain, fatigue, sleep quality, stress level, quality of life and work efficiency.

DETAILED DESCRIPTION:
Considering the importance of the workforce and possible health problems in white-collar workers, it seems rational to implement health promotion practices in accordance with the digital age. There is no study in the literature examining the effectiveness of technology-based yoga on selected health outcomes in white-collar workers. Based on this shortcoming, the aim of this study is to examine the effects of yoga exercises applied with two different technological access in white-collar employees on musculoskeletal pain, fatigue, sleep quality, stress level, quality of life and work efficiency.

ELIGIBILITY:
Inclusion Criteria:

* • Working full-time in the last 1 year in administrative, research-development, high-tech education, mind and brain power-based jobs

  * Speaks and writes Turkish
  * In order to join online sessions, participants should have internet access
  * All answers of the Physical Activity Preparation Survey should be selected as "No"

Exclusion Criteria:

* • Uncontrolled hypertension and uncontrolled arrhythmia patience

  * Individuals who have undergone percutaneous transluminal coronary angiography or have a cardiac pacemaker
  * Individuals with severe neurological disease or serious respiratory disease
  * Previous stroke, myocardial infarction
  * Individuals who have undergone amputation
  * Individuals with major musculoskeletal problems
  * Individuals with injuries involving the lower extremity in the past 6 months
  * Pregnant or planning a pregnancy within 1 year
  * Breastfeeding
  * Use of sleeping pills or medication for psychological problems and/or shift workers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
physical activity level | 8 weeks
  International Physical Activity Questionnarie -Short Form: This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.

SECONDARY OUTCOMES:
musculoskeletal pain level | 8 weeks
  Nordic Musculoskeletal Questionnaire: The questionnaire consists of four parts. In the first part, first name, last name, date of questioning, gender, date of birth, body weight, length of stature, dominant side, how many years/months has he been working in the current job and how many hours worked on average in a week are recorded. In the second part the last 12 months, individuals in nine different body regions (neck, shoulder, back, elbow, waist circumference, wrist/hand, hip/thigh, knee, and ankle/foot) with the presence of pain or discomfort experienced the pain of blocking the Activity Status is questioned. The third section nine different body areas of pain or discomfort experienced in the last 7 days individuals in the presence and in the final chapter, an individual one of these areas which, when applied to the physician because of pain or discomfort in questioned.
fatigue severity. | 8 weeks
  The Fatigue Severity Scale: It is shown as the best example among one-dimensional decimals. It consists of a total of 9 questions, and each question on the scale is scored from 1 (I don't agree at all) to 7 (I completely agree). The total score of the scale dec from 9 to 63. The fact that the total score that can be obtained from the scale is 36 or higher indicates severe fatigue.
sleep quality | 8 weeks
  Pittsburgh Sleep Quality Index: The scale evaluates the individual's sleep quality, amount of sleep and the presence of sleep disorder. There are 19 questions answered by the individual himself and 5 questions answered by the individual's roommate in the scale, which consists of 24 questions in total. However, when calculating the total score of the scale, the questions answered by the roommate are not included in the calculation. The scoring includes 18 items and 7 components: subjective sleep quality, sleep latency (delay), sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction. Each item is scored between 0-3. The total score of the scale is calculated by the sum of the scores from the seven components, and the total score ranges from 0 to 21 points. A total score of 5 or more indicates poor sleep quality.
perceived stress | 8 weeks
  Perceived Stress Index: The Perceived Stress Scale will be used to evaluate the stress level of the participants. The scale was developed to identify the source of stress and the level of perceived stress. The questions in the scale should be answered by taking into account the feelings and thoughts in the last month. It consists of 14 items in total and each item is rated with a 5-point Likert-type scale. High scores obtained from the scale indicate that the perception of stress is high.
quality of life of the participants | 8 weeks
  Short Form-36 will be used to assess the participants' quality of life. The scale developed by Corporation consists of 36 items and 8 sub-dimensions. Sub-dimensions of the scale; physical function (10 items), social function (2 items), role limitations due to physical functions (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items) and general perception of health (5 items). Each item in the scale should be answered considering the last four weeks. Instead of a single total score from the scale, each sub-dimension is scored separately. The sub-dimension score ranges from 0 to 100. 0 points indicate poor health and 100 points indicate good health.
work efficiency | 8 weeks
  Endicott Productivity at Work scale: The scale consists of 25 items and besides these items, the number of hours the individual has to work, the number of hours he has worked, and if he has worked less than necessary, the reason for this is questions. The 25 items related to work efficiency are never (0), rarely (1), sometimes (2), often (3), or almost always (4), depending on how often the individual's behavior, emotion, or attitude has been seen in the previous week. as a score. The lowest total score that can be obtained from the scale is 0 and the highest total score is 100. A high score indicates low work efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akıncı, Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No